CLINICAL TRIAL: NCT05871164
Title: Longitudinal, Prospective, French, Multicenter Cohort Study on Pancreatic Radiofrequency
Acronym: RAFPAN2
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A00247-38
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient to be treated for a tumor of the pancreas: Patient to be treated for a tumor of the pancreas by ultrasound-guided radiofrequency with a fine needle, with Indication of pancreatic radiofrequency validated in a Multidisciplinary Consultation Meeting
  Interventions: Procedure: Pancreatic radiofrequency

INTERVENTIONS:
Procedure: Pancreatic radiofrequency — Pancreatic radiofrequency is similar to a puncture under echoendoscopy. The lesion is located then punctured by transgastric or transduodenal route either using a 19 gauge needle with exchange of the stylet for a probe, or using a 19 gauge needle whose distal end of 5-10 mm corresponds to the active part, connected to a generator with an integrated cooling system.

SUMMARY:
The purpose of the study is to evaluate the oncological efficacy of pancreatic radiofrequency by the objective response rate (complete and partial responses according to RECIST 1.1.), 5 years after the end of treatment.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, open, non-randomized, non-interventional, multicenter study on ultrasound-guided radiofrequency endoscopy for the treatment of pancreatic tumours. The study will be offered prospectively to all patients in need of treatment. They will be taken care of in accordance with current practice.

The patient will be seen again 7 times after the end of the pancreatic radiofrequency (which will include one or two sessions): the follow-ups will be done according to current practice on D15 ± 7 days, M6 ± 14 days, M12 ± 1 month then annually until M60 ± 1 month.

The study consists to evaluate the oncological efficacy at 5 years of pancreatic radiofrequency delivered by means of a needle guided by ultrasound endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Patient to be treated for a pancreatic tumor by ultrasound-guided RF with a fine needle;
* Indication of pancreatic radiofrequency validated in a Multidisciplinary Consultation Meeting;
* Patient able to understand the information related to the study;
* Patient accepting study follow-up visits;
* Patient having been informed and agreeing to participate in the study.

Exclusion Criteria:

* Patient with a contraindication to radiofrequency treatment;
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 to be treated for pancreatic tumor by ultrasound-guided radiofrequency with fine needle
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Carcinological efficacy of pancreatic radiofrequency | 5 years
  The primary endpoint of the study is the oncological efficacy of pancreatic radiofrequency, which will be assessed by the objective response rate (complete and partial responses according to RECIST 1.1.), 5 years after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Toulon La Seyne, Toulon, France